CLINICAL TRIAL: NCT06453980
Title: Multimodal Investigation of Neural Plasticity Induced by Non-invasive Brain Stimulation
Brief Title: Multimodal Investigation of Neural Plasticity
Acronym: miniSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Alzheimer's Association (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Alexandru Iordan, Assistant Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00201483
Record Dates: First submitted 2024-05-17; First posted 2024-06-12 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment
Keywords: tDCS; Glutamate; MRS; fMRI; fNIRS
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Healthy controls (HC) and individuals with MCI will be randomized 1:1:1:1 to receive either sham or active stimulation (i.e., HC sham tDCS, HC active tDCS, MCI sham tDCS, MCI active tDCS) for 1 session using a blocked randomization design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- HC sham tDCS (Sham Comparator): Sham (placebo) dose of HD-tDCS treatment for 20 minutes, for 1 session.
  Interventions: Device: sham tDCS
- HC active tDCS (Experimental): 3 milliAmp dose of HD-tDCS treatment for 20 minutes, for 1 session.
  Interventions: Device: active tDCS
- MCI sham tDCS (Sham Comparator): Sham (placebo) dose of HD-tDCS treatment for 20 minutes, for 1 session.
  Interventions: Device: sham tDCS
- MCI active tDCS (Experimental): 3 milliAmp dose of HD-tDCS treatment for 20 minutes, for 1 session.
  Interventions: Device: active tDCS

INTERVENTIONS:
Device: sham tDCS — Participants will receive sham (placebo) HD-tDCS for 20 minutes, for 1 session.
  Arms: HC sham tDCS; MCI sham tDCS
Device: active tDCS — Participants will receive HD-tDCS at 3 milliAmp for 20 minutes, for 1 session.
  Arms: HC active tDCS; MCI active tDCS

SUMMARY:
This study will evaluate the effects of a form of non-invasive brain stimulation on brain functioning and memory in cognitively intact older adults (healthy controls, HC) and in those with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The goal of this study is to learn important information about the effects of weak electrical stimulation (known as high-definition transcranial direct current stimulation or HD-tDCS) on brain functioning in those with mild cognitive impairment (MCI). The findings will help determine how stimulation affects brain's activity and metabolism (in particular, the neurotransmitter glutamate). Ultimately, this information may help develop new treatments for those with Alzheimer's disease. The study will use different forms of brain imaging to see whether stimulation changes how the brain responds during a memory task. Functional magnetic resonance spectroscopy (fMRS), functional magnetic resonance imaging (fMRI), and functional near-infrared spectroscopy (fNIRS) will be used. The study also uses cognitive tests and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognition for HC and diagnosis of Mild Cognitive Impairment (MCI) for MCI participants
* Right-handedness
* Magnetic resonance compatible, criteria that also apply for high definition transcranial direct current stimulation (HD-tDCS; e.g., absence of metallic or electronic implants in the upper body or head)

Exclusion Criteria:

* History of other contributing neurological or medical conditions known to affect cognitive functioning
* Significant mental illness
* Sensory impairments that limit ability to participate
* History of alcohol or drug abuse/dependence

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in glutamate concentration (fMRS) | average on 1 week
  Analyses via fMRS using units of concentration
Changes in brain activation (fMRI) | average of 1 week
  Analyses via fMRI using units of brain activation

SECONDARY OUTCOMES:
Changes in memory performance | average of 1 week
  Analyses of memory performance indexed as percent accuracy
Changes in brain activation (fNIRS) | immediate, concurrent with tDCS
  Analyses via fNIRS using units of brain activation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Iordan, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No